CLINICAL TRIAL: NCT01706809
Title: Comparing of Different Biomarkers From Vena Rectalis Superior and Vena Cubiti in Patients Undergoing Low Anterior Resection for Rectum Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mark Ellebaek Pedersen, Medical doctor, Odense University Hospital
Other Study IDs: S-20100006; S-20100006
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biomarkeres
  Interventions: Other: blood sampels from vena rectalis superior and vena cubiti

INTERVENTIONS:
Other: blood sampels from vena rectalis superior and vena cubiti

SUMMARY:
The primary aim of the present study is to investigate different biomarkers like VEGF, EVGF and others ability to predict time to recidive and progressions free survival.

DETAILED DESCRIPTION:
Patients undergoing LAR for rectum cancer is subjected. Preoperative blood samples from vena rectalis superior and vena cubiti is collected, as well as biopsies from tumor. Preoperative and after 3 month peripheral blood samples is collected.

A total of 50 patients will be included in this study.

The study is approved by the local scientific ethical committee No. S-20100006

ELIGIBILITY:
Inclusion Criteria:

* Histological verified cancer
* The cancer must be located in rectum maximum of 15 cm.
* Age above 18

Exclusion Criteria:

* Disseminated cancer
* Perioperative radio-chemotherapy
* Laparoscopy surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing open LAR for rectum cancer is subjected.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The primary aim of the present study is to investigate different biomarkers like VEGF, EVGF and others ability to predict time to recidive and progressions free survival. | after the study is complete

CONTACTS AND LOCATIONS:
Locations (1):
- Vejle hospital, Vejle, Vejle, Denmark